CLINICAL TRIAL: NCT04524117
Title: Prediction of Vulnerable Plaque Using Coronary CT Angiography and Computational Fluid Dynamic in Acute Coronary Syndrome
Acronym: PVCFD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, MD, pHD, Director of Cardiovascular Department, Shanghai 10th People's Hospital
Other Study IDs: PVCFD
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome; Plaque, Atherosclerotic
MeSH Terms: conditions — Acute Coronary Syndrome; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A(vulnerable plaque group): Lipid plaques with fibrous cap thickness less than 65um, erosion and coronary artery dissection detected by OCT are defined as vulnerable plaque.
- Group B(stable plaque group): Lipid plaques with fibrous cap thickness more than 65um detected by OCT are defined as vulnerable plaque.

SUMMARY:
The aim of the PVCFD trial is to predict vulnerable plaque confirmed by OCT using coronary CT angiography and computational fluid dynamics in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Acute coronary syndrome（ACS）mainly includes unstable angina, non-ST-segment elevation myocardial infarction, and ST-segment elevation myocardial infarction, which is the leading cause of death around the world. The main pathophysiological feature of ACS is the rupture of vulnerable plaque, which can be recognized by coronary artery angiography (CAG), intravascular ultrasound (IVUS) and optical coherence tomography (OCT). Compared with CAG and IVUS, OCT is the best intravascular imaging technique so far. But all these examinations are invasive and expensive. Recently, coronary CT angiography derived adverse plaque characteristics (APC) and hemodynamic forces defined by computational fluid dynamics (CFD) can reflect plaque vulnerability and hemodynamic forces acting on the plaque, which are important factors in the progress of the rupture of vulnerable plaque. So, we want to explore predictive value of coronary CT angiography (CTA)and computational fluid dynamics for vulnerable plaque in ACS.

The PVCFD trial is a prospective and single center study, patients with ACS will be arranged to complete coronary CTA before CAG. OCT will be used to detect the characteristics of coronary atherosclerotic plaques confirmed by CAG. Lipid plaques with fibrous cap thickness less than 65um, erosion and coronary artery dissection are defined as vulnerable plaque. Patients will be divided into vulnerable plaque group and stable plaque group according to this. The coronary CTA images will be screened for APC and CFD analyses at core laboratories of Shanghai tenth's hospital. Lesions with diameter stenosis (DS) >30% based on coronary CTA evaluation were included for subsequent APC (low-attenuation plaque, positive remodeling, napkin-ring sign, and spotty calcification) analysis and hemodynamic forces (FFRCT,ΔFFRCT, WSS and PWS) defined by CFD. Three prediction models (Model 1: percent diameter stenosis + lesion length, Model 2: Model 1 + APC, Model 3: Model 2 + hemodynamic force) will be constructed to identify vulnerable plaque confirmed by OCT.

ELIGIBILITY:
Inclusion Criteria:

1)acute coronary syndrome was diagnosed according to universal definition of ACS; and 2) coronary CTA was completed before CAG; and 3) definitely culprit lesion can be recognized by CAG; 4) OCT was done to detect coronary atherosclerotic plaques confirmed by CAG.

Exclusion Criteria:

1) Previous history stent implantation; 2) previous history of coronary artery bypass graft surgery; 3) ACS without clear culprit lesion; 4) poor image quality of coronary CTA for APC and CFD analysis; 5) myocardial infarction secondary to other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The difference of area under curve among the three prediction models | from 1 to 72 hours
The difference of net reclassification index (NRI) and integrated discrimination improvement (IDI) among the three prediction models | from 1 to 72 hours

SECONDARY OUTCOMES:
The percentage in APC (low-attenuation plaque, positive remodeling, napkin-ring sign, and spotty calcification) between the vulnerable plaque group and stable plaque group | from 1 to 72 hours
The difference in hemodynamic parameters (FFRCT,ΔFFRCT, WSS and PWS) between the vulnerable plaque group and stable plaque group | from 1 to 72 hours
The optimal cut-off values of hemodynamic parameters (FFRCT,ΔFFRCT, WSS and PWS) to identify vulnerable plaque | from 1 to 72 hours